CLINICAL TRIAL: NCT03403946
Title: Comparison of Direct and Indirect Laryngoscopy Using C-MAC PM® With Macintosh Blade and D-Blade® in Simulated Difficult Airway
Brief Title: Macintosh and D-Blade® in Simulated Difficult Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Florian Raimann, Principal Investigator, Johann Wolfgang Goethe University Hospital
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 126/11
Record Dates: First submitted 2018-01-06; First posted 2018-01-19 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Difficult Intubation; Cervical Injury Spine
Keywords: difficult airway; carvical collar; endotracheal intubation
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All patients received the same treatment.
  1. Laryngscopy with C-MAC PM + Macintosh blade
  2. Laryngscopy with C-MAC PM + D-Blade
  3. Intubation with C-MAC PM + D-Blade
  Interventions: Device: Macintosh blade; Device: D-Blade; Device: Intubation

INTERVENTIONS:
Device: Macintosh blade — Laryngoscopy with C-MAC PM in combination with Macintosh blade
Device: D-Blade — Laryngoscopy with C-MAC PM in combination with D-Blade
Device: Intubation — Intubation with C-MAC PM in combination with D-Blade

SUMMARY:
In the presented study, our aim was to compare intubation conditions regarding the modified Cormack & Lehane score (CL) between the D-Blade® in indirect laryngoscopy or Macintosh blade in direct and indirect laryngoscopy with C-MAC PM® in a simulated setting of a difficult airway in human subjects.

DETAILED DESCRIPTION:
Patients with unexpected difficult airway requiring endotracheal intubation (ETI) remain extremely challenging for emergency physicians and intubation failure with subsequent hypoxic complications still represents the majority of cases in a recent closed claims analysis.

An incidence of major complications in airway management of 1 in 5,500 was estimated in the Fourth National Audit Project in the UK.

Therefore, our aim was to compare intubation conditions regarding the modified Cormack & Lehane score (CL) between the D-Blade® in indirect laryngoscopy or Macintosh blade in direct and indirect laryngoscopy with C-MAC PM® in a simulated setting of a difficult airway in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring general anesthesia for orthopedic surgery

Exclusion Criteria:

* known or expected difficult airway
* undergoing urgent or emergent surgery
* non-fasted
* American Society of Anesthesiology Class (ASA) IV-VI
* no consent for participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2012-08-31 (Actual)

PRIMARY OUTCOMES:
Best view of the glottic structures | 120 seconds after induction of narcosis
  Best view of the glottic structures according to the modified Cormack and Lehane (CL) scoring system

SECONDARY OUTCOMES:
Evaluate the process of Intubation using a questionnaire | Directly after successful tracheal intubation
  As a secondary endpoint, all investigators were asked to evaluate the process of ETI with the D-Blade® from grade 1 to grade 4.
  Grade 1: Uncomplicated ETI with guide rod Grade 2: Challenging ETI, readjustment or usage of BURP necessary Grade 3: ETI using a stylet Grade 4: ETI failed
Subjective assessment of satisfaction using numeric rating scale | Directly after successful tracheal intubation
  Finally, all investigators were asked for their subjective assessment from 0 = dissatisfied to 100 = fully satisfied when using the D-Blade®.

CONTACTS AND LOCATIONS:
Overall Officials: Haitham Mutlak, Dr. med., Study Director — Department of Anesthesia, Intensive Care Medicine and Pain Therapy
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raimann FJ, Dietze PE, Cuca CE, Meininger D, Kessler P, Byhahn C, Gill-Schuster D, Zacharowski K, Mutlak H. Prospective Trial to Compare Direct and Indirect Laryngoscopy Using C-MAC PM(R) with Macintosh Blade and D-Blade(R) in a Simulated Difficult Airway. Emerg Med Int. 2019 Apr 1;2019:1067473. doi: 10.1155/2019/1067473. eCollection 2019. PMID 31065384